CLINICAL TRIAL: NCT02449707
Title: Evaluation of a Lateral Window Technique Augmentation for Maxillary Sinus Lift Using Ultrasound Activated Resorbable Poly-D-L-lactide Pins in Maxillary Sinus Lift - a Split Mouth Randomized Control Trial
Brief Title: Evaluation of a Lateral Window Technique Augmentation for Maxillary Sinus Using Ultrasound Activated Pins
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Dr Sharat Pani, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FRP/2014/109
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Lateral Window Technique Augmentation for Maxillary Sinus without the use of Ultrasound activated resorbable poly-D-L-lactide pins for the stabilization of membrane. Placement of Purus® Cancellous Allograft, stabilized by Biomend ™ Collagen membrane. Cone Beam CT image of the sinus will be taken to evaluate the bone formation. Trephine Biopsy will be performed after 1 year, at the time of placement of implant to check the quality of bone formed.
  Interventions: Procedure: Lateral Window Technique Augmentation for Maxillary Sinus; Device: Purus® Cancellous Allograft; Device: Biomend; Procedure: Cone Beam CT image of the Sinus; Procedure: Trephine Biopsy
- Ultrasonic Pins (Experimental): Lateral Window Technique Augmentation for Maxillary Sinus with the use of Ultrasound activated resorbable poly-D-L-lactide pins for the stabilization of the Purus® Cancellous Allograft, and Resorb X Membrane.Cone Beam CT image of the sinus will be taken to evaluate the bone formation. Trephine Biopsy will be performed after 1 year, at the time of placement of implant to check the quality of bone formed.
  Interventions: Procedure: Lateral Window Technique Augmentation for Maxillary Sinus; Device: Ultrasound activated resorbable poly-D-L-lactide pins; Device: Purus® Cancellous Allograft; Device: Resorb X Membrane; Procedure: Cone Beam CT image of the Sinus; Procedure: Trephine Biopsy

INTERVENTIONS:
Procedure: Lateral Window Technique Augmentation for Maxillary Sinus — Maxillary sinus augmentation will be performed using the lateral window technique
Device: Ultrasound activated resorbable poly-D-L-lactide pins — The titanium membrane placed during the maxillary sinus augmentation procedure will be stabilized using ultrasound activated resorbable poly-D-L-lactide pins
  Other Names: Sonic Weld
  Arms: Ultrasonic Pins
Device: Purus® Cancellous Allograft — Allograft material placed in the sinus to acheive sinus augmentation
Device: Resorb X Membrane — The membrane placed over the graft material before placement of the ultrasound activated pins
  Arms: Ultrasonic Pins
Device: Biomend — Collagen healing membrane placed over the graft material on the side where no ultrasound activated pins are being used
  Arms: Control
Procedure: Cone Beam CT image of the Sinus — Cone beam CT will used to assess the thickness of bone formation after the placement of the graft
Procedure: Trephine Biopsy — Trephine Biopsy will be performed at the time of the placement of implant to study the quality of bone formed

SUMMARY:
Ultrasound activated pins have been used for the promotion of bone healing in combination with biodegradable membranes during bone grafting procedures. In the jaws, these pins have been successfully tested for both maxillary and mandibular ridge augmentaton. However, the usefulness of these pins in maxillary sinus lift procedures has not been tested. This study aims to use a bilateral split mouth design to compare the bone formation, healing and post-operative complications after the use of ultrasonic guided pins in a lateral window maxillary sinus augmentation procedure in comparison to lateral window maxillary sinus augmentation procedure procedure performed without the use of these pins.

DETAILED DESCRIPTION:
The study proposes to use a prospective split mouth crossover randomized control trial design to study the success of implant placement in cases with sinus lift procedures performed using the Sonic Weld® (KLS-Martin GmbH , Mulheim, Germany) ultrasound guided bone welding system with a membrane (Resorb X Membrane) on one side, and placement of Biomend collagen membrane to stabilize the graft

Patient selection:

20 patients requiring bilateral maxillary sinus lift procedure (40 procedures) will be selected from the patients reporting for implant placement to both the Riyadh Colleges of Dentistry and Pharmacy and the Riyadh Dental Center, King Saud Medical City.

Graft Placement:

Each patient will receive both the pin stabilized and the conventional graft placement procedures with standardized allografts (Purus® Cancellous Allograft?) on both sides of the maxilla. The grafts will be placed using the lateral window technique. The patients will be randomly assigned into either those who receive the pin first (Group A) or those who receive the conventional technique (using collagen membranes) first (Group B). The patients will have a one week gap between the sinus lift on the right and left sides.

Evaluations of the sinus lift procedure:

The sinus lift will be evaluated clinically radiographically and histologically using previously established criteria. Cone Beam CTs (Gallelios Comfort plus, Sirona Dental, Salzburg, Austria) will be taken preoperatively and at three month intervals to help assess the osseous outcomes of the graft.

At the end of one year the site will be evaluated clinically for the placement of implants. At the time of placement of the implant a trephine biopsy will be performed and H&E staining will be used to determine the histological outcomes of the graft procedure.

Statistical Analysis:

The paired t test will be used to compare the thickness of bone before and after the completion of the sinus lift procedure. The multiple measures paired ANOVA will be used to compare the thickness of bone at each follow up vist.

The student's t test will be used to compare the thickness of bone between the two types of sinus lift procedure.

The chi-square test will be used to compare differences (if any) in the histological patterns obtained at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Loss of upper permanent molar on both right and left side
* Require Bilateral Maxillary Sinus Augmentation
* Consent to partipate in the study

Exclusion Criteria:

* History of Diabetes Mellitus (including patients who are controlled with oral hypoglyceamic drugs)
* Uncontrolled Hypertensive patients with three consecutive diastolic readings of over 90mmHg
* History of Osteoporosis

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in bone thickness (in mm) | Change from Baseline thickness in 6 months

SECONDARY OUTCOMES:
Change in Post-operative pain - as reported on a Visual Analog Scale (VAS) | Change from baseline VAS in 6 months
Bone Quality - Measured by the type of bone observed on the trephine biopsy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bishi AlGarni, MSc, Study Chair — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia